CLINICAL TRIAL: NCT00758563
Title: Train New Examiners Via Modified Gingival Margin Plaque
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-0907-PLA-18-RR
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2008-11-20 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Fluorides; Triclosan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: Fluoride
- B (Active Comparator)
  Interventions: Drug: Triclosan/Fluoride

INTERVENTIONS:
Drug: Fluoride — Brush twice daily
  Arms: A
Drug: Triclosan/Fluoride — Brush twice daily
  Arms: B

SUMMARY:
The purpose of this study is to train new examiners while testing two commercial products using our standard one-day brushing study regimen by measuring gingival margin plaque index.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers 18-65 years of age
* Good general health
* Must sign informed consent form
* Must discontinue oral hygiene for 24-hrs.after initial appointment.
* Minimum of 20 natural uncrowned teeth (excluding third molars) must be present.
* No history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study.

Exclusion Criteria:

* Subjects unable or unwilling to sign the informed consent form.
* Medical condition which requires pre-medication prior to dental visits/procedures
* Moderate or advanced periodontal disease or heavy dental tartar (calculus).
* 2 or more decayed untreated dental sites at screening.
* Other disease of the hard or soft oral tissues.
* Impaired salivary function (e.g. Sjogren's syndrome or head and neck irradiation).
* Use of medications that can affect salivary flow
* Use of antibiotics or antimicrobial drugs within 30 days prior to study visit #1.
* Pregnant or nursing women.
* Participation in any other clinical study within 1 week prior to enrollment into this study.
* Use of tobacco products
* Subjects who must receive dental treatment during the study dates.
* Current use of Antibiotics for any purpose.
* Presence of an orthodontic appliance.
* History of allergy to common dentifrice ingredients.
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Sigal-Greene, Principal Investigator
Locations (1):
- Northampton Community College, Bethlehem, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At clinical site
Period: Overall Study
Arm/Group | Fluoride | Triclosan
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoride | Triclosan | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.3 (17.4) | 32.1 (11.5) | 33.1 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Gingival Plaque Units
Description: Scale 0 to 100% of tooth gingival margin covered by plaque. (0=no plaque, 100%=100% of the tooth's gingival margin is covered in plaque).
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fluoride | Triclosan
Number analyzed (Participants) | 7 | 8
Units on a scale | 13.38 (13.65) | 14.29 (12.25)
Statistical Analysis 1: Comparison: Fluoride vs Triclosan; Test type: Superiority or Other; p = 0.05, ANOVA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days